CLINICAL TRIAL: NCT06521502
Title: The ARDS, Pneumonia, and Sepsis (APS) Consortium: A Prospective Observational Study to Evaluate Phenotypes
Brief Title: The APS Phenotyping Study
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wesley Self, APS Consortium Coordinating Center Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 240088
Record Dates: First submitted 2024-07-16; First posted 2024-07-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: ARDS; Sepsis; Pneumonia
Keywords: acute respiratory distress syndrome; sepsis; pneumonia; phenotype; endotype; critical illness
MeSH Terms: conditions — Sepsis; Pneumonia; Respiratory Distress Syndrome; Critical Illness | interventions — Blood Specimen Collection; Urine Specimen Collection; Surveys and Questionnaires; Hand Strength; Muscle Strength

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens to be collected include blood; urine; stool; oral, nasal, and rectal swabs; heat moisture exchange (HME) filter fluid; tracheal aspirate; and non-bronchoscopic bronchoalveolar lavage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A (full study protocol - written informed consent): Cohort A is the cohort of APS study participants who have provided written informed consent for participation in the APS phenotyping study. Cohort A may participate in all study procedures in the APS phenotyping study.
  Interventions: Other: Blood collection; Other: Urine Collection; Other: Nasal, oral, and rectal swabs; Other: Stool collection; Other: Heat Moisture Exchange Filter collection; Other: Tracheal Aspirate sample collection; Procedure: Non-bronchoscopic bronchoalveolar lavage (NBBAL); Other: Surveys
- Cohort B (alteration study protocol - alteration of informed consent): Cohort B is the cohort of APS study participants who are enrolled in the study under alteration of informed consent. Cohort B will participate in a modified set of procedures which omits procedures considered greater than minimal risk.
  Interventions: Other: Blood collection; Other: Urine Collection; Other: Nasal, oral, and rectal swabs; Other: Stool collection; Other: Heat Moisture Exchange Filter collection; Other: Tracheal Aspirate sample collection
- Long-term Outcomes Cohort: The Long-term Outcomes Cohort consists of a subset of participants with written informed consent for study participation (Cohort A) who complete in-person post-hospital study assessments. These in-person study visits are scheduled at 3-, 6-, and 12-months after initial enrollment in the hospital. Interventions/exposures are denoted for this group for study procedures that are completed during an in-person post-hospital visit.
  Interventions: Other: Blood collection; Other: Nasal, oral, and rectal swabs; Other: Stool collection; Other: Short physical performance battery; Other: Hand grip strength; Other: CNS Vital Signs; Other: Muscle Ultrasound; Other: Muscle Strength; Other: Spirometry; Other: Lung Diffusion Testing (DLCO); Radiation: Chest CT Scan

INTERVENTIONS:
Other: Blood collection — Blood will be collected from a catheter ("IV") that is already in place or using a needle stick into a vein.
  Blood will be collected in hospital (Cohorts A, B) and at visits 3, 6, and 12 months following hospitalization for (Long-term Outcomes Cohort).
Other: Urine Collection — Urine will be collected through a urinary catheter that is already in place or by urinating into a cup.
  Urine will be collected in hospital only (Cohorts A, B)
  Groups: Cohort A (full study protocol - written informed consent); Cohort B (alteration study protocol - alteration of informed consent)
Other: Nasal, oral, and rectal swabs — Nasal, oral, and rectal swabs inserted into the nose, mouth, and rectum, respectively. The swabs will be rubbed inside the cavity and then removed the swab.
  Oral and nasal swabs will also be collected in hospital (Cohort A, B) and at visits 3, 6, and 12 months following hospitalization for (Long-term Outcomes Cohort). Rectal swabs will be collected in hospital only (Cohorts A, B).
Other: Stool collection — Stool will be collected either in a cup after defecation or by collecting it from a tube or bag that may already be in place that is catching stool.
  Stool will be collected in hospital (Cohorts A, B) and at visits 3, 6, and 12 months following hospitalization (Long Term Outcomes Cohort).
Other: Heat Moisture Exchange Filter collection — An HME filter is a sponge that is placed in the tubing between a patient and breathing machine. It reduces the amount of heat and moisture a patient loses when on a breathing machine. Moisture from breath is collected in this filter. The filter is changed every few hours. When the filter is changed, it will be saved to collect the moisture that it contains and run tests on it.
  HME filters will be collected in hospital on intubated patients only (Cohorts A, B).
  Groups: Cohort A (full study protocol - written informed consent); Cohort B (alteration study protocol - alteration of informed consent)
Other: Tracheal Aspirate sample collection — Patients on a breathing machine have a breathing tube in their trachea that connects their lungs to the breathing machine. A smaller tube, called a suction catheter, will be placed through the larger tube and fluid will be gently sucked out.
  Tracheal aspirate will be collected in hospital on intubated patients only (Cohorts A, B)
  Groups: Cohort A (full study protocol - written informed consent); Cohort B (alteration study protocol - alteration of informed consent)
Procedure: Non-bronchoscopic bronchoalveolar lavage (NBBAL) — The NBBAL procedure involves putting a flexible rubber tube through the breathing tube into the airway of one of the lungs. A small amount of fluid is injected into the lung and then a gentle suction is used to collect fluid. Only patients who pass a safety screen showing that they are not at high risk for complications will have the NBBAL procedure performed.
  NBBAL will be performed in hospital on intubated patients only (Cohort A)
  Groups: Cohort A (full study protocol - written informed consent)
Other: Surveys — Participants will be contacted by email, text, and /or phone to give updates about their health. These surveys will ask questions about quality of life, mental health, return to work, and re-admission to the hospital. (Cohort A)
  Groups: Cohort A (full study protocol - written informed consent)
Other: Short physical performance battery — At visits 3, 6, and 12 months following hospitalization (Long-term Outcomes Cohort)
  Chair Stand Test: For this test the participant will sit in a chair. They will then stand as quickly as possible without using their upper body to assist them.
  Balance Test: For this test the participant will stand unsupported for 10 seconds with their feet in 3 different positions.
  4-meter walk: For this test the participant will walk 4 meters as quickly as possible.
  Groups: Long-term Outcomes Cohort
Other: Hand grip strength — At visits 3, 6, and 12 months following hospitalization (Long-term Outcomes Cohort):
  The participant will squeeze a machine called a hand-held dynamometer 3 times with all their strength.
  Groups: Long-term Outcomes Cohort
Other: CNS Vital Signs — At visits 3, 6, and 12 months following hospitalization (Cohort A - Long-term Outcomes Cohort):
  The participant will sit at a computer and follow the prompts on the screen. This test takes about 45 minutes.
  Groups: Long-term Outcomes Cohort
Other: Muscle Ultrasound — At visits 3, 6, and 12 months following hospitalization (Long-term Outcomes Cohort):
  The participant will undergo ultrasound on the quadriceps muscle on the dominant side of their body.
  Groups: Long-term Outcomes Cohort
Other: Muscle Strength — At visits 3, 6, and 12 months following hospitalization (Long-term Outcomes Cohort):
  A dynamometer will be used to measure muscle strength in the dominant leg.
  Groups: Long-term Outcomes Cohort
Other: Spirometry — At a visit 12 months following hospitalization (Long-term Outcomes Cohort):
  The participant will have a clip placed on their nose and will be given a plastic mouthpiece that is connected to a machine called a spirometer. They will place their lips tightly around the mouthpiece and take in as big and deep of a breath as possible and then blow out as hard and fast as they can.
  Groups: Long-term Outcomes Cohort
Other: Lung Diffusion Testing (DLCO) — At a visit 12 months following hospitalization (Long-term Outcomes Cohort):
  The participant will have a clip on their nose. They will put their mouth over a mouthpiece that is attached to a machine. This machine will deliver a small amount of carbon dioxide when they breathe in and will also record the results of the test. They will then take a few normal breaths. Next they will inhale deeply and exhale completely. They will breathe in quickly through their mouth and hold their breath for 10 seconds or as long as they can. Then they will breathe out.
  Groups: Long-term Outcomes Cohort
Radiation: Chest CT Scan — At a visit 12 months following hospitalization (Long-term Outcomes Cohort):
  The participant will undergo a Chest Computed Tomography (CT) scan which uses special X-ray equipment to take detailed pictures of the lungs.
  Groups: Long-term Outcomes Cohort

SUMMARY:
The goal of the observational APS phenotyping study is to better understand risk factors, potential biomarkers, length and severity of illness, and recovery for adults with ARDS, pneumonia, and/ or sepsis. This study will also generate a biobank of specimens collected from these patients that will be available to investigators for future studies of ARDS, sepsis, and/or pneumonia.

DETAILED DESCRIPTION:
The APS phenotyping study will enroll hospitalized adult patients ≥18 years old who have or are at risk of developing ARDS, sepsis, or pneumonia. Participation in this study will involve collection of clinical data, completing questionnaires, and collection of samples such as blood, urine, and stool. Participants who are mechanically ventilated will also provide samples from their respiratory track. Data and samples will be collected both during and after hospitalization. Analyses to understand the mechanisms underlying ARDS, pneumonia, and sepsis will be conducted, with goals including the classification of patients with ARDS, pneumonia, and sepsis into biologically based phenotype categories and identifying new targets for future therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for enrollment, a patient must meet all the following inclusion criteria at the time of the first study-specified biospecimen collection (Time 0):

1. Age ≥ 18 years old
2. Admitted (or planned to be admitted) to an intensive care unit (ICU) or other in-patient hospital location where IV vasopressors or advanced respiratory support (invasive mechanical ventilation, non-invasive ventilation, or high flow nasal cannula) are routinely provided (referred to as an "eligible unit.")
3. Acute cardiovascular or pulmonary organ dysfunction defined by meeting at least one of the two criteria below:

   * New receipt of invasive mechanical ventilation, non-invasive ventilation, high flow nasal cannula, or supplemental oxygen at a flow rate of ≥ 6 lpm for acute hypoxemia.

     a. Patients who use chronic oxygen therapy are eligible to participate if they are receiving at least 6 lpm higher than their baseline oxygen requirement (e.g., a patient on 3 lpm O2 at baseline is eligible if they require ≥9 lpm for hypoxemia) or are started on advanced respiratory support (invasive mechanical ventilation, non- invasive ventilation, or high flow nasal cannula).
   * Receipt of intravenous infusion of a vasopressor medication for at least one hour.
4. Acute cardiovascular or pulmonary organ dysfunction (inclusion criterion #3) is attributed to an acute inflammatory condition, including but not limited to any of the following:

   * Any infection including pneumonia.
   * Aspiration pneumonitis.
   * Pancreatitis.
   * Auto-inflammatory condition such as:

     1. Hemophagocytic lymphohistiocytosis.
     2. Suspected acute rheumatologic or auto-immune disease with pulmonary or cardiovascular manifestations.
     3. Suspected cryptogenic organizing pneumonia presenting acutely.
     4. Suspected diffuse alveolar hemorrhage.
     5. Suspected acute anaphylaxis.
     6. Suspected acute pulmonary drug toxicity.

Exclusion Criteria:

To be eligible for enrollment, a patient must not meet any of the following exclusion criteria at the time of the first study-specified biospecimen collection (Time 0):

1. Patient/legally authorized representative (LAR) declines participation.
2. Acute cardiovascular or pulmonary organ dysfunction (inclusion criterion #3) has been present for > 48 hours.
3. Patient has been in an eligible unit (inclusion criterion #2) for more than 120 hours (five days).
4. Patient is no longer expected to meet the acute cardiovascular or pulmonary organ dysfunction inclusion criterion (inclusion criterion #3) 24 hours after enrollment.
5. Patient desires comfort measures only.
6. Patient is a prisoner.
7. Patient had out-of-hospital cardiac arrest leading to this hospitalization.
8. Residence immediately before this hospitalization in a long-term acute care facility.
9. Presence of tracheostomy for respiratory failure.
10. Home invasive mechanical ventilation or non-invasive ventilation (except patients with non-invasive ventilation prescribed as a treatment for a sleep disorder may participate).
11. Suspected cause of the patient's acute cardiovascular and/or pulmonary dysfunction (inclusion criterion #3) is an alternative condition (not ARDS, pneumonia, or sepsis), including but not limited to the list below:

    * Drug overdose (without aspiration, lung injury, pneumonia, or infection).
    * Trauma (without aspiration, pneumonia, or infection).
    * Chronic lung disease without suspected infection, aspiration, or inflammation.
    * Asthma, chronic obstructive pulmonary disease (COPD), sarcoidosis, interstitial lung disease, neuromuscular respiratory failure.
    * Status epilepticus.
    * Acute pulmonary embolism.
    * Acute decompensated heart failure.
    * Diabetic ketoacidosis.
    * Acute stroke or intracranial hemorrhage.
    * Acute bleeding (GI bleeding, post-procedural bleeding, hemolysis).
    * Cytokine release syndrome due to chemotherapy.
12. Inability or unwillingness to complete study-specified blood draws, for example, due to local policies about hemoglobin thresholds for research blood draws.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls hospitalized adult patients ≥18 years who have or are at high risk of developing ARDS, pneumonia, and/or sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
ARDS, pneumonia, and sepsis classification | Through day 7
  Classification of critically ill adults into disease categories based on published paradigms, including the Berlin Criteria for ARDS, Sepsis-3 criteria for sepsis, and Centers for Disease Control and Prevention (CDC) criteria for pneumonia.

SECONDARY OUTCOMES:
Death | 28 days, 3 months, 6 months, 12 months
  All-cause mortality

OTHER OUTCOMES:
Invasive ventilator free days | In-hospital through day 28
  Days alive and free of invasive mechanical ventilation through day 28
Ventilatory support free days | In-hospital through day 28
  Days alive and free of invasive mechanical ventilation (IMV), non-invasive ventilation (NIV), and high flow nasal cannula (HFNC) through day 28
Vasopressor free days | In-hospital through day 28
  Days alive and free of vasopressor use through day 28
New kidney replacement therapy free days | In-hospital through day 28
  Days alive and free of new kidney replacement free days through day 28
Organ support free days | In-hospital through day 28
  Days alive and free of IMV, NIV, HFNC, vasopressors, and new kidney replacement therapy
Coma and delirium free days | In hospital through day 7
  Days alive and free of coma and delirium (defined by confusion assessment method (CAM)-ICU and Richmond Agitation Sedation Scale (RASS score) through day 7
Oxygen free days | In hospital through day 28
  Days alive and free of new supplemental oxygen therapy through day 28
Hospital free days | In hospital through day 28
  Days alive and out of the hospital through day 28
ICU free days | In hospital through day 28
  Days alive and out of the ICU through day 28
Acute kidney injury (AKI) | In hospital through day 28
  AKI defined by creatinine criteria from Kidney Disease Improving Global Outcomes (KDIGO)
Major adverse kidney events (MAKE) | In-hospital through day 28
  Death, new kidney replacement therapy, or persistent doubling of serum creatinine
Extracorporeal membrane oxygenation (ECMO) | In-hospital through day 28
  New receipt of ECMO therapy
Sequential Organ Failure Assessment (SOFA) score | Through day 7
  Organ dysfunction scoring system that assesses the performance of 6 organ systems (respiratory, cardiovascular, hepatic, renal, coagulation, and neurological). Score range is 0 to 24. A higher score indicates greater (worse) organ dysfunction.
Central Nervous System (CNS) vital signs score | 3, 6, 12 months
  CNS vital signs is a computer-based neurocognitive assessment that evaluates memory, psychomotor speed, reaction time, complex attention and cognitive flexibility. The summary score is called the Neurocognitive Index. Scoring produces a relative score for the individual relative to the American normative sample controlled for age; mean score is 100; the standard deviation is 15; higher scores represent better neurocognitive function.
Short Physical Performance Battery Protocol | 3, 6, 12 months
  Physical performance assessment
Handgrip strength | 3, 6, 12 months
  Physical strength assessment
Quadriceps muscle ultrasound | 3, 6, 12 months
  Physical muscle fitness assessment
Pulmonary spirometry, including forced vital capacity (FVC), and forced expiratory volume in 1 second (FEV1). | 12 months
  FVC is the volume of air that can be forcibly exhaled after full inspiration, measured in liters. FEV1 is the volume of air that can be forcibly exhaled in 1 second after full inspiration, measured in liters.
Diffusing capacity for carbon monoxide (DLCO) | 12 months
  Lung function assessment
EuroQol-5 Dimension-5 Level (EQ-5D-5L) quality of life assessment | 3, 6, 12 months
  A tool to measure health related quality of life. A score of 1 indicates the best possible health state and a score <0 is the worst possible health state.
Impact of Event Scale (IES)-6 | 3, 6, 12 months
  PTSD assessment scored out of 4, with a score of ≥ 1.75 denoting likely PTSD
Hospital Anxiety and Depression Scale (HADS) | 3, 6, 12 months
  A fourteen-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.
Modified Medical Research Council (mMRC) dyspnea score | 3, 6, 12 months
  The mMRC scale is a self-assessment tool used to measure the level of impairment caused by breathlessness during daily activities, rated on a scale from 0 (no breathlessness) to 4 (severe limitation).
Clinical frailty scale | 3, 6, 12 months
  A nine-point scale based on clinical evaluation of mobility, energy, physical activity, and function. Higher scores indicate increased frailty.
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 | 3, 6, 12 months
  A tool that measures how a health condition affects a person's ability to function in everyday life. Scored from 0-100 where 0 indicates no disability and 100 indicates full disability.
Return to work | 3, 6, 12 months
  Assessment of returning to work after critical illness
Financial toxicity | 3, 6, 12 months
  Assessment of financial stress after critical illness
Housing instability | 3, 6, 12 months
  Assessment of housing after critical illness

CONTACTS AND LOCATIONS:
Overall Officials: Wesley H. Self, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (18):
- United States (18):
  - Fresno Community Hospital and Medical Center, Fresno, California
  - Stanford University, Palo Alto, California
  - San Francisco General Hospital, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Denver, Colorado
  - Denver Health and Hospital Authority, Denver, Colorado
  - National Jewish Health, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins Univeristy, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
During conduct of the APS Consortium study procedures, data, biospecimens, and radiographic images will be collected by enrolling sites and transmitted to the APS Consortium Coordinating Center at Vanderbilt University Medical Center. Data and biospecimens will be organized and catalogued at the coordinating center. Additionally, the coordinating center will periodically transmit data and biospecimens to repositories managed by the National Heart, Lung, and Blood Institute (NHLBI) -- BioData Catalyst (data repository) and BioLINCC (biospecimen repository).
  During the period of performance for the APS Consortium, requests for data and/or biospecimens for use in ancillary studies will be reviewed for approval by the APS Steering Committee.
  After the completion of the APS Consortium period of performance, requests for data and/or biospecimens for use in ancillary studies will be governed by NHLBI through the BioData Catalyst and BioLINCC programs.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The first large subset of APS data and biospecimens is anticipated to be available for distribution no earlier than the first quarter of calendar year 2026. The full cohort of data and biospecimens will be available in 2028.
Access Criteria: Requests for use of biospecimens and/or data will be reviewed by the APS Consortium Steering Committee through the end of the program. After the program has completed, requests will be reviewed by the US National Heart, Lung, and Blood Institute (NHLBI).
URL: http://apsconsortium.org

REFERENCES:
- [Background] Semler MW, Bernard GR, Aaron SD, Angus DC, Biros MH, Brower RG, Calfee CS, Colantuoni EA, Ferguson ND, Gong MN, Hopkins RO, Hough CL, Iwashyna TJ, Levy BD, Martin TR, Matthay MA, Mizgerd JP, Moss M, Needham DM, Self WH, Seymour CW, Stapleton RD, Thompson BT, Wunderink RG, Aggarwal NR, Reineck LA. Identifying Clinical Research Priorities in Adult Pulmonary and Critical Care. NHLBI Working Group Report. Am J Respir Crit Care Med. 2020 Aug 15;202(4):511-523. doi: 10.1164/rccm.201908-1595WS. PMID 32150460
- See also: Notice of Funding Opportunity (NOFO) for APS Consortium — http://grants.nih.gov/grants/guide/rfa-files/RFA-HL-23-001.html